CLINICAL TRIAL: NCT01480037
Title: Genetic and Physiological Aspects of Oxidative Profile in Sleep and Well-succeed Aging
Status: Completed | Type: Observational
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Diego Robles Mazzotti, Diego Robles Mazzotti, Associação Fundo de Incentivo à Pesquisa
Other Study IDs: LONG-2011
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Aging; Without Mention of Psychosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples collected for DNA and RNA extraction, as well as for laboratory examinations
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Elderly: Individuals between 60 and 70 years-old
- Long-lived: Individuals above 85 years-old
- Young: Individuals between 20 and 30 years-old

SUMMARY:
The present study proposes the characterization of sleep patterns of healthy young adults, elderly individuals and individuals above 85 years old, using polysomnographic recordings, in order to clarify the importance of sleep in longevity. Furthermore, this study intends to analyze the oxidative stress-related gene expression in peripheral blood of the three studied groups, using the Superarray - RT2 Profiler" PCR Array System. After the identification of genes whose expression pattern among groups suggest a more specific role in longevity, the mechanisms of gene expression regulation, including DNA methylation patterns and microRNA expression, as well as the possible genomic sources of variation in these genes will be investigated. In addition, the oldest individual (105 years-old) will have his whole genome sequenced using next-generation sequencing technology, in order to identify rare variants associated with longevity. Subsequently, the effect of the polymorphisms and rare variants identified will be confirmed in an expanded sample constituted of individuals with various age-ranges. The study will provide a better characterization of molecular and physiological mechanisms involved in longevity, hoping to contribute to the development of more advanced clinical tools, capable to offer a better quality of life for the elderly.

DETAILED DESCRIPTION:
In the last decades, the increase in life expectancy highlights the world population aging as an irreversible process. The oxidative stress hypothesis of aging suggests that accumulation of oxidative damage during lifespan may be related to loss of cellular functions, a process normally associated with senescence. However, it has been proposed that individuals who live longer in a successful manner tend to be more adapted against aging physiological changes. Sleep is essential in maintaining health and well-being. Growing evidence suggests interrelationships between oxidative stress and sleep, while the latter is an important mechanism involved in redox balance maintenance. Therefore, the present study proposes the characterization of sleep patterns of healthy young adults, elderly individuals and individuals above 85 years old, using polysomnographic recordings, in order to clarify the importance of sleep in longevity. Furthermore, this study intends to analyze the oxidative stress-related gene expression in peripheral blood of the three studied groups, using the Superarray - RT2 Profiler" PCR Array System. After the identification of genes whose expression pattern among groups suggest a more specific role in longevity, the mechanisms of gene expression regulation, including DNA methylation patterns and microRNA expression, as well as the possible genomic sources of variation in these genes will be investigated. In addition, the oldest individual (105 years-old) will have his whole genome sequenced using next-generation sequencing technology, in order to identify rare variants associated with longevity. Subsequently, the effect of the polymorphisms and rare variants identified will be confirmed in an expanded sample constituted of individuals with various age-ranges. The study will provide a better characterization of molecular and physiological mechanisms involved in longevity, hoping to contribute to the development of more advanced clinical tools, capable to offer a better quality of life for the elderly.

ELIGIBILITY:
Inclusion Criteria:

* men aged between 20-30 years-old,
* 60-70 years-old and above 90 years-old

Exclusion Criteria:

* Uncontrolled chronic disease (cancer, cardiopathy, type 2 diabetes)
* neurological and/or psychiatric antecedents

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of São Paulo city, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Polysomnography parameters | 1 night
Gene expression data | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Tufik, MD PhD, Study Director — Associação Fundo de Incentivo à Pesquisa
Locations (1):
- Associação Fundo de Incentivo à Pesquisa, São Paulo, São Paulo, Brazil